CLINICAL TRIAL: NCT06062576
Title: Clinical Efficacy Observation and Mechanism Study of Yunnan Baiyao in Different Stages of Diabetic Foot
Brief Title: Clinical Observation and Mechanism Study of Yunnan Baiyao in Different Stages of Diabetic Foot
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Peking University Third Hospital (Other)
Responsible Party: Principal Investigator, Long Zhang, Professor, Peking University Third Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Long2023-DFU-YunnanBaiyao
Record Dates: First submitted 2023-09-25; First posted 2023-10-02 (Actual); Last update posted 2024-06-25 (Actual); Status verified 2024-06

CONDITIONS: Diabetic Foot; Therapeutics
Keywords: Diabetic Foot; Therapeutics
MeSH Terms: conditions — Diabetic Foot | interventions — yunnan baiyao

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (6):
- control group 1 (No Intervention): The optimal clinical treatment scheme was used to treat the wound of progressive infection period patients for 2 weeks
- powder group 1 (Experimental): On the basis of the optimal clinical treatment scheme, Yunnan Baiyao powder was used to treat the wound of progressive infection period patients for 2 weeks
  Interventions: Drug: Yunnan Baiyao
- ointment group 1 (Experimental): On the basis of the optimal clinical treatment scheme, Yunnan Baiyao ointment was used to treat the wound of progressive infection period patients for 2 weeks
  Interventions: Drug: Yunnan Baiyao
- control group 2 (No Intervention): The optimal clinical treatment scheme was used to treat the wound of granulation period patients for 2 weeks
- powder group 2 (Experimental): On the basis of the optimal clinical treatment scheme, Yunnan Baiyao powder was used to treat the wound of granulation period patients for 2 weeks
  Interventions: Drug: Yunnan Baiyao
- ointment group 2 (Experimental): On the basis of the optimal clinical treatment scheme, Yunnan Baiyao ointment was used to treat the wound of granulation period patients for 2 weeks
  Interventions: Drug: Yunnan Baiyao

INTERVENTIONS:
Drug: Yunnan Baiyao — On the basis of the optimal clinical treatment scheme, Yunnan Baiyao powder or ointment was used to treat the wound for 2 weeks
  Arms: ointment group 1; ointment group 2; powder group 1; powder group 2

SUMMARY:
Yunnan Baiyao has been treating all kinds of wounds for 120 years, but the evidence of Evidence-based medicine that is truly convincing is insufficient, making its best application method unclear. This study explored the possible indications and use methods of Yunnan Baiyao in different stages of Diabetic foot, and obtained Evidence-based medicine evidence of clinical efficacy. Obtain the discarded tissues of Diabetic foot patients in the treatment and control groups of Yunnan Baiyao after wound debridement, conduct Transcriptome (BulkRNA seq) analysis and detection on the wound tissues, and analyze the related signal pathways and functional genes with significant differences, to help clarify the possible treatment targets of Yunnan Baiyao.

ELIGIBILITY:
Inclusion Criteria:

1. The age of the subjects is 18-80 years old;
2. Diagnose diabetes according to WHO standards;
3. Diagnosis of Diabetic foot;
4. Confirmed as one of the stages of infection progression and granulation growth;
5. Voluntarily participate in this study and sign an informed consent form.

Exclusion Criteria:

1. Severe diseases such as acute myocardial infarction, heart failure, hepatitis, shock, and respiratory failure have not been corrected yet;
2. Blood glucose is out of control, Glucose test#Fasting blood sugar>15mmol /L, Glycated hemoglobin>12%;
3. There is active bleeding inside the wound, and routine basic treatment plans cannot be implemented;
4. Serum albumin<20g/L; Hemoglobin<60g/L; Platelets<50 × 109/L;
5. Late stage subjects with malignant tumors;
6. Active period of autoimmune diseases;
7. Have a history of allergy to Yunnan Baiyao;
8. The subject is unable to cooperate or has mental disorders;
9. According to the judgment of the researcher, the subject has a clear reason that cannot be removed and affects wound healing, which is not suitable for this study or cannot comply with the requirements of this study.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2023-12-01 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2025-06-30 (Estimated)

PRIMARY OUTCOMES:
2-week reduction rate of wound area | 2 weeks
  Difference in wound area before and after treatment

CONTACTS AND LOCATIONS:
Locations (1):
- Peking University 3rd Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No